CLINICAL TRIAL: NCT04419779
Title: A Prospective, Randomized, Double-Blind, Sham-Controlled, Multi-Center, Pivotal Study to Evaluate the Efficacy and Safety of Duodenal Mucosal Resurfacing Using the Revita® System in Subjects With Type 2 Diabetes With Inadequate Glycemic Control
Brief Title: Evaluation of the Efficacy and Safety of DMR Using the Revita® in Subjects With Inadequately Controlled Type 2 Diabetes
Acronym: REVITALIZE 1
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment pause
Sponsor: Fractyl Health Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-00044
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Revita System; Duodenal Mucosal Resurfacing; Insulin-Dependent Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Duodenal Mucosal Resurfacing (DMR) (Active Comparator): Duodenal Mucosal Resurfacing (DMR) treatment will include hydrothermal ablation of the duodenal muscosa in an upper endoscopic procedure in patients with inadequately controlled type 2 diabetes.
  Interventions: Device: Duodenal Mucosal Resurfacing (DMR)
- Duodenal Mucosal Resurfacing Sham (Sham) (Sham Comparator): Duodenal Mucosal Resurfacing Sham (Sham) treatment will include an upper endoscopic procedure similar to DMR treatment without hydrothermal ablation of the duodenal mucosa in patients with inadequately controlled type 2 diabetes.
  Interventions: Device: Duodenal Mucosal Resurfacing (Sham)

INTERVENTIONS:
Device: Duodenal Mucosal Resurfacing (DMR) — The Fractyl DMR Procedure utilizes the Revita® Catheter to perform hydrothermal ablation of the duodenum. The Catheter is delivered trans-orally over a guide-wire to first inject saline to lift the sub-mucosal space, followed by an ablation of the duodenal mucosa. Subjects who receive the DMR treatment are followed for 48 weeks post treatment.
  Arms: Duodenal Mucosal Resurfacing (DMR)
Device: Duodenal Mucosal Resurfacing (Sham) — The Sham procedure consists of placing the Revita® Catheter as described above into the duodenum for a minimum of 30 minutes and then removing it from the patient. Subjects who receive the Sham procedure are followed for 48 weeks post treatment and are offered cross over to undergo the DMR procedure at 48 weeks and are followed for further 48 weeks post treatment. Sham subjects who choose not to cross over are discontinued from the study.
  Arms: Duodenal Mucosal Resurfacing Sham (Sham)

SUMMARY:
The Revita® system is being investigated to assess the efficacy of DMR versus Sham on improvement in Glycemic, Hepatic and Cardiovascular endpoints for patients with Type 2 Diabetes who are inadequately controlled on one or more glucose lowering agents. The purpose of this study is to demonstrate the efficacy and safety of the Fractyl DMR Procedure using the Revita® System compared to a sham. Subjects randomized to the DMR procedure will be followed per protocol till 48 weeks post treatment. Subjects in the Sham treatment arm will be offered cross over to receive the DMR treatment at 48 weeks and will be followed per protocol for 48 weeks post treatment.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria for inclusion in the study:

1. Males and non-pregnant non-lactating females
2. Age between 21 and 70 years (both inclusive)
3. Subjects on at least one glucose lowering agent (GLA) with no changes in GLA medications or dosing for at least 12 weeks prior to the screening visit

   Permitted GLAs include:
   * Metformin,
   * GLP-1 RA including dual peptide agonists and related molecules (e.g., GLP-1/GIP RA),
   * DPP-4i,
   * TZDs,
   * SGLT2is,
   * SUs,
   * Meglitinides,
   * Insulin (basal or basal combined with short-acting), up to a total of 100 units daily
4. HbA1c of 7.5%-10% (both inclusive)
5. BMI >24 to ≤40 kg/m2
6. WOCBP should have a negative urine beta hCG pregnancy test and must agree to use two of the established contraceptive methods throughout the study duration
7. Able to sign an ICF and comply with study requirements

Exclusion Criteria

Subjects who meet any of the following exclusion criteria are not allowed to be included in the study:

1. FPG ≥270 mg/dL
2. Known case of absolute insulin deficiency as indicated by clinical assessment or a fasting plasma C-peptide of <0.6 ng/mL
3. Subjects on any other class of glucose-lowering agents other than GLAs listed in inclusion criteria Any drugs or concomitant medications (e.g., psychoactive drugs such as carbamazepine phenobarbital; sympathomimetics such as ephedrine corticosteroids; anabolic steroids and male sex hormones such as testosterone) that can interfere with glucose metabolism (refer to prohibited medication on Appendix D: Eligibility Criteria Checklist)
4. Recurrent or severe urinary tract or genital mycotic infections or history of GU infection within 4 weeks prior to informed consent, for those subjects on SGLT-2
5. ALT or AST >3 times upper limit of normal (ULN) for the reference range, as determined by the central laboratory at screening visit. Patients with NAFLD are eligible if their ALT level is ≤3.0 times the ULN.
6. Use of an investigational drug within 1 month or 5 half-lives (whichever is longer) before screening
7. Diagnosed with type 1 diabetes or with a recent history of DKA within one year prior to screening
8. Ketosis-prone T2D
9. Known diabetes related non-healing ulcers or amputations (with the exception of a finger or toe amputation occurring > 1 year prior to screening.
10. History of more than 1 severe hypoglycemia episode or hypoglycemia unawareness within the last 6 months
11. Clinically significant hypoglycemia occurring during the run-in period, defined as a) 2 or more glucose alert values of ≤70 mg/dL (3.9 mmol/L) unless a clear, correctable, precipitating factor can be identified; b) clinically significant hypoglycemia with self-monitored or laboratory plasma glucose level <54 mg/dL (3.0 mmol/L); or c) severe hypoglycemic episode requiring third party assistance
12. Known intestinal autoimmune disease including celiac disease, ulcerative colitis, Crohn's disease, lupus erythematosus, scleroderma, or other autoimmune connective tissue disorder that affects the small intestine
13. Secondary hypothyroidism or inadequately controlled primary hypothyroidism (thyroid stimulating hormone [TSH] value outside the normal range at screening as determined by the central laboratory).
14. Known thyroid cancer or hyperthyroidism with treatment within the past 12 months or inadequately controlled hyperthyroidism (TSH value outside the normal range at screening as determined by the central laboratory).
15. An uncontrolled endocrine condition such as multiple endocrine neoplasia (except T2D)
16. Known structural or functional disorder of the esophagus including any swallowing disorder, esophageal chest pain disorders, drug-refractory esophageal reflux symptoms, or active and uncontrolled gastroesophageal reflux disease (GERD) (defined as Los Angeles Grade C or D esophagitis)
17. Known structural or functional disorder of the stomach including active gastric ulcer, chronic gastritis, gastric varices, hiatal hernia (a large hiatal hernia or type II and higher paraoesophageal hernia), cancer, or any other disorder of the stomach
18. Previous GI surgery that could affect the ability to treat the duodenum such as subjects who have had a Billroth 2, Roux-en-Y gastric bypass, gastric sleeve, or other similar procedures or conditions
19. Known history of chronic pancreatitis or a recent history of acute pancreatitis within the past year
20. Presence of acute or chronic active hepatitis B or C (except if hepatitis C is cured) or cirrhosis, hepatic decompensation/acute liver disease during the last 6 months, or alcoholic or autoimmune chronic hepatitis
21. Symptomatic gallstones, symptomatic kidney stones, or acute cholecystitis
22. Clinically active systemic infection
23. Known immunocompromised status including but not limited to individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months; have clinically significant leukopenia; are positive for the human immunodeficiency virus (HIV); are on potential immunosuppressants; or individuals whose immune status makes the subject a poor candidate for clinical trial participation in the opinion of the investigator
24. Known active malignancy or partial remission from clinically significant malignancy within the past 5 years (except basal or squamous cell skin cancer, carcinoma in situ, those who received curative treatment and are in complete remission for 5 years, or if the subject is confirmed as cancer free)
25. Known active coagulopathy or current upper gastro-intestinal bleeding conditions such as ulcers, gastric varices, strictures, or congenital or acquired intestinal telangiectasia
26. Known cases of sickle cell anemia, thalassemia, or conditions that affect red blood cell (RBC) turnover such as a recent blood transfusion within 90 days. Current persistent anemia, defined as hemoglobin <10g/dL
27. Use of anticoagulation therapy (e.g., warfarin, coumadin, or novel oral anticoagulants [NOACs]) or anti-platelet agents (e.g., thienopyridine) which cannot be discontinued for 5-7 days or 2 drug half-lives before the procedure
28. Use of systemic glucocorticoids (excluding topical or ophthalmic applications or inhaled forms) for more than 10 consecutive days within 90 days prior to screening
29. Use of non-GLA drugs known to affect GI motility (e.g., metoclopramide)
30. Known moderate to severe chronic kidney disease (CKD) with an estimated glomerular filtration rate (eGFR) of <45 mL/min/1.73m2 (estimated by Modification of Diet in Renal Disease [MDRD]), end-stage renal failure, or on dialysis
31. History of myocardial infarction, stroke, transient ischemic attack, coronary artery intervention, CHF exacerbation, or any other major cardiac event requiring hospitalization within the last 6 months prior to screening or any cardiac history that would deem subject not eligible for anesthesia (unless documented clearance by cardiologist and/or treating endoscopy team)
32. History of new or worsening signs or symptoms of coronary heart disease (CHD) within the last 3 months
33. Known case of severe peripheral vascular disease, defined as AMA Criteria Class 1 or greater75 (Appendix 19.8)
34. Known case of symptomatic heart failure with reduced ejection fraction (NYHA Class II-IV) requiring pharmacologic therapy to control symptoms
35. Clinically significant electrocardiogram (ECG) findings such as new clinically significant arrhythmia, ST segment changes, or other conduction disturbances that increase risk of heart disease and require intervention as determined by the investigator
36. Subjects who are at risk of pancreatitis, particularly those with a recent fasting triglyceride value of >600 mg/dL within the past 3 months
37. Actively participating in a weight-loss program and currently not in the maintenance phase
38. General contraindications to deep or conscious sedation, general anesthesia, high risk as determined by anesthesiologist (e.g., ASA score 4 or higher), or contraindications to upper GI endoscopy
39. History of substance use disorder based on the DSM-5 criteria76 within the last 12 months (American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition).
40. Use of weight loss medication such as Meridia, Xenical, over-the-counter weight-loss medications, or other prescribed medications used specifically for the purpose of weight loss
41. Use of dietary supplements or herbal preparations that may have unknown effects on glycemic control or risk of bleeding
42. Participating in another ongoing clinical trial of an investigational drug or device
43. History of non-adherence to treatment in the previous 6 months, as determined by the investigator based on patient history, HbA1c value, or drug accountability
44. Any other mental or physical condition which, in the opinion of the investigator, makes the subject a poor candidate for clinical-trial participation. Physical conditions assessed via endoscopy prior to participant study enrollment at visit 4 include, but not limited to:

    1. Active and uncontrolled gastroesophageal reflux disease (GERD) defined as Los Angeles Grade C or D esophagitis
    2. Abnormalities of the GI tract preventing endoscopic access to the duodenum
    3. Anatomic abnormalities in the duodenum that would preclude the completion of the DMR procedure, including tortuous anatomy
    4. Malignancy newly diagnosed by endoscopy
    5. Upper GI conditions (esophageal, gastric, or intestinal) such as clinically significant ulcers, polyps, varices, strictures, congenital or acquired intestinal telangiectasia, or other conditions listed under exclusion criteria
45. Unwilling or unable to comply with study visits and other study procedures as required per protocol
46. Recovered from severe COVID-19 infection (requiring hospitalization) but with persistent long COVID-19 symptoms (i.e., the individual has not recovered for several weeks or months since the start of symptoms that were suggestive of COVID-19, irrespective if the individual was tested or not)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate superiority of Revita DMR to sham in improving glycemic control | Baseline to Week 24
  Change from baseline in HbA1c at Week 24

SECONDARY OUTCOMES:
Demonstrate superiority of Revita DMR to sham in achieving target HbA1c at 24 weeks | Baseline to Week 24
  The proportion of subjects who achieve an HbA1c of ≤7.0% at Week 24
Demonstrate superiority of Revita DMR to sham in fasting glucose at 24 weeks | Baseline to Week 24
  Change from baseline in fasting plasma glucose (FPG) at Week 24
Demonstrate superiority of Revita DMR to sham in weight loss at 24 weeks | Baseline to Week 24
  Percentage of total body weight loss (%TBWL) from baseline at Week 24
To demonstrate superiority of Revita DMR to sham in elimination of insulin use at 24 weeks in those subjects on insulin at baseline | Baseline to Week 24
  4. The proportion of subjects who discontinued insulin at Week 24 in those subjects on insulin at baseline

CONTACTS AND LOCATIONS:
Locations (58):
- United States (51):
  - Helios CR, Inc, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Angel City Research , Inc., Los Angeles, California
  - UCLA Health, Los Angeles, California
  - Care Access Santa Clarita, Newhall, California
  - Hoag Hospital, Newport Beach, California
  - Stanford University Medical Center, Redwood City, California
  - Mills Peninsula Health Center, San Mateo, California
  - Northeast Research Institute, Llc, Fleming Island, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Advent Health Orlando, Orlando, Florida
  - Synexus Research, Orlando, Florida
  - Northwestern Unviersity, Evanston, Illinois
  - AHN - Avon, Avon, Indiana
  - Investigators Research Group, Brownsburg, Indiana
  - AHN- Franklin, Franklin, Indiana
  - AHN - Greenfield, Greenfield, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - AHN - Muncie, Muncie, Indiana
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Alcanza Clinical Research, LLC, Methuen, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - IMA Clinical Research St. Louis, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Endocrine Associates of West Village, Long Island City, New York
  - NYU Langone Gastroenterology Associates, New York, New York
  - Synexus Clinical Research, New York, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - M3 Wake Research, Raleigh, North Carolina
  - AcellaCare Salisbury, Salisbury, North Carolina
  - AcellaCare Piedmont, Statesville, North Carolina
  - AcellaCare Wilmington, Wilmington, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Preferred PCP - Pittsburgh, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Care Access Warwick, Warwick, Rhode Island
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Biopharma Informatic, Llc, Houston, Texas
  - Simcare Medical Research, Llc., Sugar Land, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels, Belgium
- University College Dublin, Dublin, Ireland
- Italy Gemelli, Roma, Italy
- Universiteit Van Amsterdam Academisch Medisch Centrum, Amsterdam, Netherlands
- University Hospital Zurich, Zurich, Switzerland
- United Kingdom (2):
  - Cleveland Clinic London, London, England
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No